CLINICAL TRIAL: NCT01297114
Title: Imaging of Cognition, Learning, and Memory in Aging
Status: Completed | Type: Observational
Sponsor: Yaakov Stern (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor-Investigator, Yaakov Stern, Professor of Neuropsychology, Columbia University
Organization: Columbia University (Other)
Other Study IDs: AAAB0596; R01AG026158 (NIH)
Record Dates: First submitted 2011-02-14; First posted 2011-02-16 (Estimated); Last update posted 2017-11-01 (Actual); Status verified 2017-10

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — 4-(N-methylamino)-4'-(2-(2-(2-fluoroethoxy)ethoxy)ethoxy)stilbene

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Whole blood (frozen)
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Participants aged 60-70: Participants age 60-70 will receive Florbetaben PET tracer to identify presence of amyloid burden.
  Interventions: Drug: Florbetaben
- Participants aged 20-30: Younger participants will not undergo PET scanning that will be studied with other methods.

INTERVENTIONS:
Drug: Florbetaben — This is a purely observational study. Results of the Florbetaben PET scan will be correlated with other observations.
  Other Names: F-18 BAY
  Groups: Participants aged 60-70

SUMMARY:
This investigation is designed to study how the brain functions when it is performing explicit memory tasks, and furthermore how the brain systems supporting performance on these tests change as a function of aging. Implicit memory tasks may be distinguished from explicit memory tests in that explicit memory characterizes the directed or intentional recollection of previously learned information or events. In contrast, implicit (or nonconscious) memory is expressed in the facilitation of performance on some task or judgment on a stimulus owing to a prior presentation of that stimulus, without any necessary conscious awareness of the prior presentation. The investigators propose to use functional Magnetic resonance Imaging (fMRI) to measure brain activity during the performance of carefully designed explicit memory tasks. Comparison of brain activity during the different test conditions will provide information about the brain areas that are involved in mediating specific aspects of performance. Both older and younger individuals will be tested in order to understand age related changes in the brain activity. In order to examine the interactions between participants' differential levels of amyloid burden and their performance on cognitive tasks and fMRI neural activation, the investigators also propose PET imaging of older participants.

DETAILED DESCRIPTION:
The basic approach to measuring the brain activity associated with a given cognitive process (or processes) is as follows: It is known that increases in brain neuronal activity are associated with local increases in energy metabolism. Under normal circumstances, increases in brain metabolism lead to local changes in blood oxygenation in venules and larger veins. This change in blood oxygenation can be detected imaging methods which are sensitive to the differences in magnetic state between oxygenated and deoxygenated hemoglobin.

The ultimate benefit of this research is to better understand how changes in both performance and the brain organization underlying that performance are affected by aging.

ELIGIBILITY:
Inclusion Criteria:

* Aged 20-30 or 60-70
* Residing near Columbia University Medical Center
* Must be willing and able to participate

Exclusion Criteria:

* Have a contraindication to PET (e.g, metallic implants, pacemaker, claustrophobia, or cannot lie flat for one hour)
* Pregnancy
* Lactating Women
* Current, past, or anticipated exposure to radiation
* Significant active physical illness

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects will be recruited from ads placed in local newspapers and notices posted in the vicinity of Columbia University, the Columbia Presbyterian Medical Center, and in local senior centers that provide written consent for notice placement. We will also utilize a market mailing approach. Letters will be sent to appropriately aged potential subjects randomly selected from commercial lists. Additional elderly subjects will be recruited from the Sergievsky Joint Database. Informed consent will be elicited from all subjects.
Sampling Method: Probability Sample
Enrollment: 294 (Actual)
Dates: Start 2011-03; Primary Completion 2017-10-01 (Actual); Study Completion 2017-10-01 (Actual)

PRIMARY OUTCOMES:
Cognition as measured with cognitive evaluations | cross sectional
  We will assess the relationship between the presence of amyloid and cognition as measured with standard cognitive and neuropsychological tests

CONTACTS AND LOCATIONS:
Overall Officials: Yaakov Stern, PhD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data could be shared based on NIH regulations
Time Frame: Study data will be available within 1 year
Access Criteria: We will be sharing de-identified data with a consortium that is aggregating studies that have employed amyloid PET tracers

REFERENCES:
- [Background] Oh H, Steffener J, Razlighi QR, Habeck C, Stern Y. beta-Amyloid Deposition Is Associated with Decreased Right Prefrontal Activation during Task Switching among Cognitively Normal Elderly. J Neurosci. 2016 Feb 10;36(6):1962-70. doi: 10.1523/JNEUROSCI.3266-15.2016. PMID 26865619
- [Background] Oh H, Steffener J, Razlighi QR, Habeck C, Liu D, Gazes Y, Janicki S, Stern Y. Abeta-related hyperactivation in frontoparietal control regions in cognitively normal elderly. Neurobiol Aging. 2015 Dec;36(12):3247-3254. doi: 10.1016/j.neurobiolaging.2015.08.016. Epub 2015 Aug 24. PMID 26382734